CLINICAL TRIAL: NCT03790813
Title: Informative Tools to Optimize Neoadjuvant Therapy in ER Positive, HER2 Negative Breast Cancers
Acronym: ER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: Genomic Health®, Inc. (Industry)
Responsible Party: Principal Investigator, Stephen Chia, Chair- British Columbia Breast Tumour Group, British Columbia Cancer Agency
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H18-02581
Record Dates: First submitted 2018-11-30; First posted 2019-01-02 (Actual); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eligible patients (Experimental)
  Interventions: Diagnostic Test: Intervention 1; Diagnostic Test: Intervention 2

INTERVENTIONS:
Diagnostic Test: Intervention 1 — Ki-67 and Oncotype DX® will be performed on the baseline core biopsy specimen prior to initiation of neoadjuvant systemic therapy.
Diagnostic Test: Intervention 2 — MRI will be performed prior to initiation of neoadjuvant systemic therapy and at the end of treatment.

SUMMARY:
This study evaluates the addition of Ki-67, Oncotype DX and MRI in the treatment of early stage breast cancer with neoadjuvant treatment. All enrolled patients will have Ki-67 and Oncotype AND/OR an MRI before and after surgery.

DETAILED DESCRIPTION:
Based on what is known about the treatment of breast cancer, there are occasional advantages to giving treatment before surgery. Some of these advantages can include shrinking a large breast cancer to facilitate surgery, shrinking a breast cancer to allow breast conservation (avoid a mastectomy), and evaluating how effective a treatment is in real-time, based on its effect on the breast cancer.

When recommending treatment with hormone therapy and/or chemotherapy, doctors take into consideration all the characteristics of a breast cancer. Over recent years, is has been recognized that additional tests can help predict the behavior of a cancer and predict the possible benefit of hormone therapy and/or chemotherapy. Because there is no way to identify exactly who benefits from chemotherapy, many patients receive chemotherapy when they might not need it.

This study involves the use of 2 separate tests. The first is called Ki-67 and is done using a piece of tumour that is taken during a needle biopsy. The second, called the Oncotype DX, is made by Genomic Health, Inc, located in Redwood, CA, USA. This test also uses a piece of tumour that was retrieved during a needle biopsy. The pieces will be tested in a specialized laboratory that can measure the levels of a specific set of genes in the tumour. The laboratory that performs this test (Redwood, CA, USA) has been certified by federal and state agencies in the United States to perform the test (called Oncotype DX). The results of the test are turned into a score (called Recurrence Score) that has been used for patients receiving treatment after surgery, but has not yet been used when treatment is given before surgery.

The standard practice for this type of cancer is for the patient and their doctor to decide whether they should receive chemotherapy in addition to hormone therapy or to take hormone therapy alone, prior to surgery. The Ki-67 is inconsistently used in British Columbia prior to surgery, but may be used routinely in other centers. Usually, the Oncotype DX test is not available to aid in this decision outside of a research study.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be between the ages (inclusive) of 18-89.
2. Patient has adequate performance status (PS ECOG 0,1 or Karnofsky performance status ≥70) and is a medically fit candidate for treatment of their cancer with systemic chemotherapy and/or hormonal therapy with no contra-indications to both systemic therapy options.
3. Patient is medically fit enough to be a surgical candidate.
4. Patient must be able to give informed consent directly or through the assistance of an interpreter.
5. Pathological confirmation of breast cancer by core biopsy.
6. Ductal or lobular breast cancer.
7. Breast cancer with a primary tumour (clinically selected T2-T4) OR clinically node positive.
8. Breast cancer is clinically palpable either in the breast, axilla or other nodal site.
9. ER positive by IHC (Allred >=4).
10. Her2Neu negative by IHC (0 or 1+) or FISH by current ASCO/CAP guidelines.

Exclusion Criteria:

1. Patient is a male with breast cancer.
2. Patients have ER negative tumors (ER-) by local or central BCCA assessment.
3. Patients have HER2 positive tumors by local or central BCCA assessment.
4. Patients have known metastatic breast cancer or develop metastatic disease prior to surgery.
5. Patients are unable to give consent or understand written language.
6. Patients with poor performance status (ECOG 2-4) in whom consideration of neoadjuvant chemotherapy OR hormonal therapy would be contraindicated.
7. Patients who are not fit enough to be a surgical candidate.
8. Pregnant women in whom consideration of neoadjuvant chemotherapy or neoadjuvant hormonal therapy would be contraindicated.
9. Patients who receive less than 2 weeks of neoadjuvant systemic therapy.
10. Patients who have not undergone surgical resection 12 months after enrollment.

For intervention 1 only:

1. Patients with tumors that on GHI central pathological review appears inadequate for the Oncotype DX® assay.
2. Patients with tumors that on BCCA pathological review appears inadequate for Ki-67 immunohistochemistry.

For intervention 2 only:

1. Patients with a pacemaker or contra-indication to MRI.

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2019-01-07 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of neoajduvant Ki-67 and Oncotype DX, defined as >=75% enrollment rate for all screened patients | 1 month
  • Technical feasibility of obtaining Ki-67 and Oncotype DX assay from a core biopsy sample in >= 75% of samples tested, prior to the initiation of systemic treatment.
Turnaround time of Ki-67 and Oncotype DX, defined as time from patient consent to date results are obtained | 1 month
  * Turnaround time will be defined as:
  * Time from patient consent to reporting of the Ki-67 and Oncotype DX
Feasibility of MRI prior to neoadjuvant systemic treatment, defined as >=75% of patients who receive an MRI before the start of neoadjuvant treatment | 6 months
  • Practical feasibility of obtaining serial MRIs with the existing means, resources and booking circumstances in >=75% of cases prior to the initiation of systemic therapy and surgical resection
Turnaround time of MRI prior to neoadjuvant systemic treatment, defined as time from patient consent to date of 1st MRI | 6 months
  Turnaround time will be defined as:
  • Time from patient consent to pre-treatment (baseline) MRI

SECONDARY OUTCOMES:
Correlation of Ki-67 and Oncotype DX to each other and to the outcome of neoadjuvant systemic treatment. | 6 months
  To characterize how the results of the Ki-67 Oncotype DX assay relate to the outcome of neoadjuvant systemic treatment and whether the results correlate to each other (Ki-67 and Oncotype DX).
Predictive association of Ki-67 and Oncotype to invasive locoregional or systemic relapse | 5 years
  • Time from study enrollment to the development of invasive locoregional or systemic breast cancer.
Predictive association of Ki-67 and Oncotype to overall survival | 5 years
  • Time from enrollment to death from any cause.
Impact of serial MRI on changes to surgical planning | 6 months
  Changes from original to final surgical plan.
Correlation of serial MRI to clinical and pathological response | 6 months
  Characterize how the results of serial MRIs affect surgical planning and how the radiological response relates to clinical response and pathological response.
Patient reported outcomes assessed by questionnaire | 6 months
  Patient reported outcomes assessed with a questionnaire exploring decisional conflict.
  9 questions are asked of patients regarding the MRI results and its impact on decision making. The scale is a 5 point scale, ranging from strongly disagree (1) to strongly agree (5). Results will be reported qualitatively.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Chia, MD, Principal Investigator — BCCA

IPD SHARING:
Plan to Share IPD: No